CLINICAL TRIAL: NCT00607672
Title: The RAS, Fibrinolysis and Cardiopulmonary Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Mias Pretorius, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 051170; HL 085740-01
Record Dates: First submitted 2008-02-04; First posted 2008-02-06 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Artery Disease; Angiotensin Converting Enzyme; Angiotensin Receptor Blockers; Cardiopulmonary Bypass; Fibrinolysis; Inflammation
Keywords: Angiotensin Converting Enzyme; Angiotensin Receptor Blockers; Cardiopulmonary Bypass; Fibrinolysis; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — Ramipril; candesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Patients are randomized to placebo prior to surgery
  Interventions: Drug: Placebo
- 2 (Active Comparator): Patients are randomized to Ramipril prior to surgery
  Interventions: Drug: Ramipril
- 3 (Active Comparator): Patients are randomized to Candesartan (ARB) prior to surgery
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1
Drug: Ramipril — Ramipril 2.5mg day 1 and 2 and then 5mg/d thereafter
  Arms: 2
Drug: Candesartan — Candesartan 16mg/d
  Arms: 3

SUMMARY:
Each year over a million patients worldwide undergo cardiac surgery requiring cardiopulmonary bypass (CPB).1 CPB is associated with significant morbidity including hemodynamic instability, the transfusion of allogenic blood products, and inflammation. Blood product transfusion increases mortality after cardiac surgery. Enhanced fibrinolysis contributes to increased blood product transfusion requirements in the perioperative period. CPB activates the kallikrein-kinin system (KKS), leading to increased bradykinin concentrations. Bradykinin, acting through its B2 receptor, stimulates the release of nitric oxide, inflammatory cytokines and tissue-type plasminogen activator (t-PA). Based on data indicating that angiotensin-converting enzyme (ACE) inhibitors reduce mortality in patients with coronary artery disease, many patients undergoing CPB are taking ACE inhibitors. While interruption of the renin-angiotensin system (RAS) reduces inflammation in response to CPB, ACE inhibitors also potentiate the effects of bradykinin and may augment B2-mediated change in fibrinolytic balance and inflammation. In contrast, angiotensin II type 1 receptor antagonism does not potentiate bradykinin and does not inhibit bradykinin metabolism.

Studies in animals suggest that bradykinin receptor antagonism inhibits reperfusion-induced increases in vascular permeability and neutrophil recruitment.A randomized, placebo controlled clinical trial of a bradykinin B2 receptor antagonist demonstrated some effect on survival in patients with systemic inflammatory response syndrome and gram-negative sepsis. In addition, we and others have shown bradykinin B2 receptor antagonism reduces vascular t-PA release during ACE inhibition. The current proposal derives from data from our laboratory and others elucidating the role of the KKS in the inflammatory, hypotensive and fibrinolytic response to CPB. Specifically, we have found that CPB activates the KKS and that ACE inhibition and smoking further increases bradykinin concentrations. During CPB, bradykinin concentrations correlate inversely with mean arterial pressure and directly with t-PA. Moreover, we have found that bradykinin receptor antagonism attenuates protamine-related hypotension following CPB. The current proposal tests the central hypothesis that the fibrinolytic and inflammatory response to cardiopulmonary bypass differ during angiotensin-converting enzyme inhibition and angiotensin II type 1 receptor antagonism.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Subjects, 18 to 80 years of age, scheduled for elective cardiac surgery requiring CPB
2. For female subjects, the following conditions must be met:

postmenopausal for at least 1 year, or status-post surgical sterilization, or if of childbearing potential, utilizing adequate birth control and willing to undergo urine beta-hcg testing prior to drug treatment and on every study day

Exclusion Criteria:

1. Left ventricle ejection fraction less than 30%
2. History of ACE inhibitor-induced angioedema
3. Hypotension (systolic blood pressure <100 mmHg and evidence of hypoperfusion)
4. Hyperkalemia (baseline potassium >5.0 mEq/L)
5. Inability to discontinue current ACE inhibitor or AT1 receptor antagonist.
6. Emergency surgery
7. Impaired renal function (serum creatinine >1.6 mg/dl)
8. Pregnancy
9. Breast-feeding
10. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
11. History of alcohol or drug abuse
12. Treatment with any investigational drug in the 1 month preceding the study
13. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
14. Inability to comply with the protocol, e.g. uncooperative attitude and unlikelihood of completing the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-08; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mias Pretorius, MBChB, MSc, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - TN Valley Healthcare System, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Billings FT 4th, Balaguer JM, C Y, Wright P, Petracek MR, Byrne JG, Brown NJ, Pretorius M. Comparative effects of angiotensin receptor blockade and ACE inhibition on the fibrinolytic and inflammatory responses to cardiopulmonary bypass. Clin Pharmacol Ther. 2012 Jun;91(6):1065-73. doi: 10.1038/clpt.2011.356. PMID 22549281
- [Derived] Gamboa JL, Pretorius M, Sprinkel KC, Brown NJ, Ikizler TA. Angiotensin converting enzyme inhibition increases ADMA concentration in patients on maintenance hemodialysis--a randomized cross-over study. BMC Nephrol. 2015 Oct 22;16:167. doi: 10.1186/s12882-015-0162-x. PMID 26494370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients scheduled for elective cardiac surgery requiring cardiopulmonary bypass were recruited from the Vanderbilt surgery clinic between 2006 and 2011.
Pre-assignment Details: Patients were excluded after enrollment if they met exclusion criteria, if surgery was canceled or if the patient changed his mind.
Groups:
- Placebo: Patients are randomized to placebo prior to surgery
- Ramipril (ACEI): Ramipril 2.5mg day 1 and 2 and then 5mg/d thereafter
- Candesartan (ARB): Patients are randomized to Candesartan 16mg/d (ARB) prior to surgery.
Period: Overall Study
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Started | 32 | 27 | 27
Completed | 28 | 24 | 22
Not Completed | 4 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB) | Total
Number analyzed (Participants) | 28 | 24 | 22 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 8 | 32
  >=65 years | 15 | 13 | 14 | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 66.14 (11.24) | 64.38 (10.35) | 67.05 (8.14) | 65.84 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 12 | 43
  Male | 9 | 12 | 10 | 31
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 22 | 74

OUTCOME MEASURES:

1. Primary Outcome: Tissue-type Plasminogen Activator (t-PA) Antigen Response
Description: To compare the effects of angiotensin II type I (AT1) receptor antagonism or angiotensin-converting enzyme (ACE) inhibition versus placebo on the fibrinolytic responses to cardiopulmonary bypass (CPB) as measured by t-PA antigen response
Time Frame: From the start of surgery until postoperative day 2
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Placebo: Placebo group
- Ramipril (ACEI): Angiotensin-converting enzyme group
- Candesartan (ARB): Angiotensin receptor blocker group
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
ng/mL
  Pre CPB | 14.36 (1.45) | 14.05 (1.86) | 11.97 (1.03)
  60min of CPB | 27.65 (3.39) | 36.67 (7.26) | 24.89 (2.96)
  Post surgery | 34.56 (3.35) | 41.11 (3.37) | 31.47 (2.61)
  Postoperative day 1 | 20.25 (2.03) | 17.10 (1.38) | 15.75 (1.32)
  Postoperative day 2 | 16.56 (1.87) | 12.49 (0.93) | 12.89 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.28, Mixed Models Analysis

2. Primary Outcome: Plasminogen Activator Inhibitor-1 (PAI-1) Response
Description: To compare the effects of AT1 receptor antagonism or ACE inhibition versus placebo on the fibrinolytic responses to CPB as measured by PAI-1 response
Time Frame: From the start of surgery until postoperative day 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
ng/mL
  Pre CPB | 15.14 (1.42) | 16.25 (2.70) | 18.28 (2.91)
  60min of CPB | 20.43 (1.63) | 19.41 (1.98) | 24.19 (3.84)
  Post surgery | 39.69 (3.78) | 41.62 (5.89) | 49.10 (7.32)
  Postoperative day 1 | 31.83 (4.47) | 26.27 (4.50) | 21.70 (2.75)
  Postoperative day 2 | 21.59 (3.77) | 17.33 (3.77) | 13.4 (1.55)
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.84, Mixed Models Analysis

3. Secondary Outcome: Blood Loss
Description: Blood loss over 24 hours as measured by chest tube output
Time Frame: First 24 hours after arrival in the intensive care unit
Measure: Mean (Standard Error); unit: mL
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
mL | 437 (35) | 470 (59) | 511 (119)
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.67, Kruskal-Wallis

4. Secondary Outcome: Re-exploration for Bleeding
Description: The percentage of patients that were taken back to the operating room for re-exploration because of bleeding
Time Frame: From arrival in intensive care unit until discharge from hospital
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
percentage of patients | 3.6 | 8.3 | 4.5
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.73, Chi-squared

5. Secondary Outcome: Blood Product Transfusion Requirement
Description: Percentage of patients that received blood product transfusion
Time Frame: From the start of surgery until discharge from hospital
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
percentage of patients
  Packed red blood cells | 67.9 | 62.5 | 2.7
  Plasma | 60.7 | 29.2 | 31.8
  Platelets | 46.4 | 29.2 | 22.7
  Cryoprecipitate | 7.1 | 4.2 | 4.5
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.04, Chi-squared — For plasma transfusion comparison. Ramipril and Candesartan versus placebo

6. Secondary Outcome: Vasopressor Drug Use
Time Frame: From the end of cardiopulmonary bypass until arrival in intensive care unit
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
percentage of patients
  Dobutamine | 35.7 | 29.2 | 27.3
  Mlrinone | 25.0 | 25.0 | 22.7
  Norepinephrine | 85.7 | 79.2 | 95.5
  Epinephrine | 7.1 | 4.3 | 13.6
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.27, Chi-squared — Comparison for norepinephrine use

7. Secondary Outcome: New Onset Atrial Fibrillation
Description: New onset atrial fibrillation based on electrocardiogram (ECG) rhythm strips with a duration longer than 10 seconds
Time Frame: From arrival in intensive care unit until discharge from hospital
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
percentage of patients | 17.9 | 16.7 | 27.3
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.62, Chi-squared

8. Secondary Outcome: Acute Kidney Injury
Description: Acute kidney injury (AKI) was defined according to Acute Kidney Injury Network (AKIN) criteria,specifically any increase in subject serum creatinine concentration of 50% or 0.3 mg/dL (26.5 umol/L) within 72 hours of surgery.
Time Frame: From the start of surgery until postoperative day 3
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
percentage of patients | 28.6 | 23.8 | 36.4
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.51, Chi-squared

9. Secondary Outcome: Stroke
Description: New onset neurological deficit with a duration of longer than 24 hours
Time Frame: From arrival in intensive care unit until discharge from hospital
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
percentage of patients | 7.1 | 4.2 | 4.5
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.87, Chi-squared

10. Secondary Outcome: Length of Hospital Stay
Time Frame: From the start of surgery until discharge from hospital
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
days | 7.7 (0.5) | 6.3 (0.6) | 8.1 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.04, Kruskal-Wallis

11. Primary Outcome: Interleukin-6 (IL-6) Response
Description: To compare the effects of AT1 receptor antagonism or ACE inhibition versus placebo on the inflammatory response to CPB as measured by IL-6
Time Frame: From the start of surgery until postoperative day 2
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
pg/mL
  Pre CPB | 6.29 (1.25) | 9.33 (3.25) | 6.44 (1.20)
  Post surgery | 116.04 (28.19) | 167.51 (35.64) | 144.76 (29.52)
  Postoperative day 1 | 224.96 (63.26) | 172.65 (68.93) | 218.16 (68.47)
  Postoperative day 2 | 166.96 (28.79) | 144.67 (46.41) | 243.72 (117.65)
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.69, Mixed Models Analysis

12. Primary Outcome: Interleukin-8 (IL-8) Response
Description: To compare the effects of AT1 receptor antagonism or ACE inhibition versus placebo on the inflammatory response to CPB as measured by IL-8
Time Frame: From the start of surgery until postoperative day 2
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
pg/mL
  Pre CPB | 16.18 (3.77) | 11.86 (1.42) | 13.38 (2.19)
  Post surgery | 66.44 (15.06) | 80.07 (20.28) | 76.76 (18.90)
  Postoperative day 1 | 46.18 (8.90) | 37.39 (6.04) | 37.11 (4.44)
  Postoperative day 2 | 34.39 (5.55) | 28.06 (5.28) | 37.77 (5.43)
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.97, Mixed Models Analysis

13. Primary Outcome: Interleukin-10 (IL-10) Response
Description: To compare the effects of AT1 receptor antagonism or ACE inhibition versus placebo on the inflammatory response to CPB as measured by the IL-10 response
Time Frame: From the start of surgery until postoperative day 2
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Number analyzed (Participants) | 28 | 24 | 22
pg/mL
  Pre CPB | 4.45 (0.47) | 5.36 (0.80) | 4.21 (0.61)
  Post surgery | 461.90 (84.64) | 815.74 (273.29) | 749.56 (199.31)
  Postoperative day 1 | 30.70 (6.91) | 26.89 (4.64) | 22.55 (3.04)
  Postoperative day 2 | 16.74 (3.09) | 14.59 (3.16) | 14.26 (2.13)
Statistical Analysis 1: Comparison: Placebo vs Ramipril (ACEI) vs Candesartan (ARB); Test type: Superiority or Other; p = 0.46, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: The patients were followed from the day of surgery until discharge from hospital, an average of 8 days
Arm/Group | Placebo | Ramipril (ACEI) | Candesartan (ARB)
Serious Adverse Events (participants affected / at risk) | 2/28 | 1/24 | 2/22
Other Adverse Events (participants affected / at risk) | 11/28 | 10/24 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | Ramipril (ACEI) (N=24) | Candesartan (ARB) (N=22)
Stroke (Nervous system disorders) | 2 | 1 | 1
In-hospital mortality (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | Ramipril (ACEI) (N=24) | Candesartan (ARB) (N=22)
Acute kidney injury (Renal and urinary disorders) | 8 | 5 | 8 — Acute kidney injury (AKI) was defined according to Acute Kidney Injury Network (AKIN) criteria, specifically any increase in subject serum creatinine concentration of 50% or 0.3 mg/dL (26.5 umol/L) within 72 hours of surgery.
New onset atrial fibrillation (Cardiac disorders) | 5 | 4 | 6 — Patient with pre-existing AF were excluded
Re-exploration (General disorders) | 1 | 2 | 1

LIMITATIONS AND CAVEATS:
We cannot exclude the possibility that our results may have been different if we studied a homogenous surgery population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No